CLINICAL TRIAL: NCT02947191
Title: The Safety and Efficacy Assessment of Collagen Membrane Combined With Human Umbilical Cord Mesenchymal Stem Cells (HUC-MSCs) Transplantation in Patients With Nasal Septum Perforation
Brief Title: Collagen Membrane Combined With HUC-MSCs Transplantation in Patients With Nasal Septum Perforation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAS-XDA-NSP/IGDB
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2016-10

CONDITIONS: Chronic Nasal Septum Perforation

ARMS (1):
- Collagen membrane + HUC-MSCs (Experimental)
  Interventions: Biological: Collagen membrane + HUC-MSCs

INTERVENTIONS:
Biological: Collagen membrane + HUC-MSCs — After separating bilateral nasal septum mucosas via septum reconstruction incision under endoscopy, the clinical grade HUC-MSCs combined with collagen membrane will be transplanted between the bilateral nasal septum mucosas and fixed. The patients will be treated with antibiotics for 1 week, and with naristillae menthae compositae, mucus promoting agent and other drugs for improving microcirculation for 1 month.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of collagen membrane combined with human clinical grade umbilical cord mesenchymal stem cells(HUC-MSCs) transplantation in patients with chronic nasal septum perforation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with nasal septum perforation area less than 1cm², and requires minimally-invasive treatment.
2. Male or female, 18-45 years old.
3. Ability and willingness to regular visit to hospital and follow up during the protocol Procedures.

Exclusion Criteria:

1. Cystic fibrosis, immotile cilia syndrome and other genetic diseases.
2. Syphilis, leprosy, tuberculosis and other specific infections.
3. Severe Sinusitis.
4. Autoimmune diseases or long term treatment with corticosteroids.
5. Alzheimer's disease.
6. Systemic diseases (e.g.,hypertension, diabetes and so on).
7. Previous history of nasal cancer or after receiving radiotherapy.
8. Drug abuse.
9. History of mental illness.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The change of integrity of nasal septum assessed by endoscopic examination | baseline, 1,2,3,4,8,12 weeks after surgery

SECONDARY OUTCOMES:
The change of nasal mucosal physiology assessed by olfactory test | baseline, 12 weeks after surgery
The change of nasal mucosal physiology assessed by nasal mucociliary clearance time (MCT) | baseline, 12 weeks after surgery
The change of nasal airway resistance assessed by rhinomanometry | baseline, 12 weeks after surgery
The change of nasal obstruction assessed by acoustic rhinometry | baseline, 12 weeks after surgery
The change of nasal obstructive symptom assessed by visual analogue scale (VAS) | baseline, 12 weeks after surgery
The change of nasal symptom severity assessed by total nasal symptom score (TNSS) | baseline, 12 weeks after surgery
Change from baseline in computed tomography (CT) | baseline, 12 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China